CLINICAL TRIAL: NCT01799096
Title: Effects of the Sugar Sucrose on Bodyweight and Energy Intake Over 28 Days in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Principal Investigator, Richard Hammersley, Professor of Health Psychology, University of Hull
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MRRH003
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Sucrose; Aspartame

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (Experimental): Receives sucrose
  Interventions: Dietary Supplement: Sucrose
- Aspartame (Placebo Comparator): Receives Aspartame sweetened drinks
  Interventions: Dietary Supplement: Aspartame

INTERVENTIONS:
Dietary Supplement: Sucrose — Sucrose in carbonated soft drinks (4 x250ml total1800 kJ per day)
  Other Names: Irn Bru
  Arms: Sucrose
Dietary Supplement: Aspartame — Intensely sweetened soft drink (no energy content)
  Other Names: Diet Irn Bru
  Arms: Aspartame

SUMMARY:
This study partially replicates two previous studies with normal weight women, and overweight women. Both found that women could compensate for sucrose added to the diet in carbonated soft drinks (4 x250ml total1800 kJ per day) when it was given blind over a period of 4 weeks. The hypothesis is that this applies also to obese women, who will not gain weight, increase overall energy intake in the diet, or eat differently whilst consuming sucrose. 42 participants shall be randomly assigned to either be given carbonated drinks that contain sucrose, or drinks that are artificially sweetened.

ELIGIBILITY:
Inclusion Criteria:

* Female
* BMI 30-35 kg/m²
* at least one period of dietary restriction of 4 weeks or more in the last 24 months

Exclusion Criteria:

* dislike of popular sweet carbonated drinks
* dieting during the last month
* history of diabetes
* having an eating disorder
* depression,
* being a smoker
* pregnant
* lactating,
* wearing a pacemaker
* currently taking medication for mood or thyroid disorders

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline | 4 weeks

SECONDARY OUTCOMES:
Mean daily dietary intake estimated from unweighed food diaries | 4 weeks

OTHER OUTCOMES:
Rated Mood | 4 weeks
  Mood was assessed 4 times per day over the study period

REFERENCES:
- [Derived] Reid M, Hammersley R, Duffy M, Ballantyne C. Effects on obese women of the sugar sucrose added to the diet over 28 d: a quasi-randomised, single-blind, controlled trial. Br J Nutr. 2014 Feb;111(3):563-70. doi: 10.1017/S0007114513002687. Epub 2013 Oct 29. PMID 24164779